CLINICAL TRIAL: NCT01826734
Title: Lacrimal Sac Dacryoliths (86 Samples): Chemical and Mineralogic Analyses
Brief Title: Analysis of 86 Dacryoliths at the University Hospital Ostrava
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Responsible Party: Sponsor
Other Study IDs: FNO-ENT-Dacryoliths
Record Dates: First submitted 2013-03-22; First posted 2013-04-08 (Estimated); Last update posted 2016-09-05 (Estimated); Status verified 2016-09

CONDITIONS: Lacrimal Apparatus Diseases; Lacrimal Duct Obstruction
Keywords: dacryolith; dacryocystorhinostomy; composition; chemical analysis; infrared spectrometry; scanning electron microscopy; elemental analysis
MeSH Terms: conditions — Lacrimal Apparatus Diseases; Lacrimal Duct Obstruction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Dacryolits during the DCR procedure.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with dacryolits: The study population consisted of patients following a dacryolit extraction procedure. The extraction procedure was not a part of this study.

SUMMARY:
Background Because dacryoliths occur at low frequency, few studies have focused on their composition.

The investigators aimed to present findings from morphological, chemical, and mineralogic analysis of 86 dacryoliths.

Methods The team studied 86 dacryoliths obtained during 832 dacryocystorhinostomies (DCR) performed for postsaccal obstruction. The samples were analyzed with atomic infrared spectrometry (80 samples), amino acid analysis (17 samples), scanning electron microscopy, and an electron microprobe with an energy dispersive detector (7 samples).

DETAILED DESCRIPTION:
INTRODUCTION It is not unusual to find a stone in the lacrimal sac during dacryocystorhinostomy (DCR). Although patients with dacryolithiasis often have a history of long-term intermittent epiphora, lacrimal sac distention, and/or partial obstruction of the nasolacrimal duct (NLD), dacryoliths are often only detected during DCR. The incidence of dacryoliths in the lacrimal sac of patients that undergo DCR ranges from 6.0-18.0%; however, the incidence of dacryoliths has not been evaluated in the general population. Unfortunately, most published studies on dacryoliths have included quite a small number of samples.

Canalicular concretions have long been associated with canaliculitis caused by actinomycotic infection. However, despite recent, significant progress, an understanding of the pathophysiology of lacrimal sac dacryoliths is still missing. Several predisposing factors have been suggested to contribute to the mechanism that gives rise to dacryolith formation. These factors include age (under 50 years old), sex (increased frequency in females), cigarette smoking, and previous occurrence of chronic dacryocystitis and primary acquired nasolacrimal duct obstruction (PANDO). Recent analyses have shown that dacryolith development may be related to lacrimal sac epithelial and NLD production of a broad spectrum of mucins and expression of two peptide members of the trefoil factor family (TFF), TFF1 and TFF3. Because dacryoliths occur at low frequency, few studies have focused on their composition.

In this study, the authors aimed to present findings from morphological, chemical, and mineralogic analysis of 86 dacryoliths.

MATERIALS AND METHODS A total of 967 primary EDCRs were performed at the Department of Otorhinolaryngology of the University Hospital of Ostrava and at the Department of Otorhinolaryngology of the Frydek-Mistek City Hospital between 1994 and April 2012. Only EDCRs performed for postsaccal stenosis/obstruction (832 procedures) were included in the study. Exclusion criteria were presaccal obstruction treatment, revision EDCRs, and incomplete follow-ups.

The study was performed in accordance with the Declaration of Helsinki, Good Clinical Practice, and applicable regulatory requirements. Written consent was obtained from all patients before the initiation of surgery and dacryolith analysis.

Among the group of 832 EDCRs, 86 stones of the lacrimal sac (dacryoliths) were found, including 61/86 (70.9%) in women and 25/86 (29.1%) in men. Clinical information was obtained from patient medical records, including the involved side, the etiology of the nasolacrimal duct (NLD) obstruction, the outcome of EDCR at one year after surgery, the size of the dacryolith, and data from dacryolith analysis. The investigators also performed infrared spectrometry, amino acid analysis, and imaging and morphological analyses with a scanning electronic microscope. The association with cigarette smoking was not examined.

Infrared spectroscopy The authors examined the dacryoliths with Fourier transform infrared spectrometry (FTIR; IMPACT 410, fy Nicolet) and a tableting method with potassium bromide (KBr). Evaluations were performed with OMNIC software, and the obtained spectra were compared with a library of spectra from kidney stones.

Amino acids analysis Proteins in the samples (≤ 20 mg) were hydrolyzed with hydrochloric acid [1,2]. Then, 1 mL of distilled water was added, the solution was filtered, then evaporated at 90 ºC under nitrogen, and the residue was dissolved in 2 mL of 1% aqueous NaOH. An aliquot (~0.5 mg of the initial sample) was transferred to another tube, the volume adjusted to ± 100 µL with 1% NaOH, and a derivatization was performed with ethyl chloroformate (4). Next, gas chromatography in tandem with mass spectrometry with a 7890A and MSD5975C (Agilent) was performed, equipped with a 30-m, VF-17ms capillary column (0.25 mm × 0.15 μm; CP8981 from HPST, Praque). Samples were run at temperatures ramped from 60 to 300 ºC at a rate of 6 ºC /min; split injection (10:1) was employed. Electron impact (EI) mass spectrometry detection at 70 eV was performed at temperatures of 230 ºC for the ion source, 250 ºC for the transfer line, and 150 ºC for the quad. We performed full-scan analyses with a helium-carrier gas flow of 1.2 mL/min.

Imaging and morphological analysis Morphological analyses were performed with a scanning electron microscope (QUANTA FEG 450, FEI Company, WA, USA). An electron microprobe with an energy dispersive detector (EDS) was used for the elemental analysis of the organic matrix of the stone and for the analysis of fine inorganic particulates in the stone.

Statistical analysis For statistical analysis, binomial confidence intervals (CI) for the success rates at the 95% CI were calculated. The two-sample t-test and X2 test were used to evaluate differences in age, sex, and surgical success between groups I and II; p<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age
* patients complaining of lacrimation
* patients following an extraction of a dacryolith

Exclusion Criteria:

* not signing the Informed Consent
* high risk of surgery (ASA IV)
* presaccal obstruction treatment
* revision EDCRs
* incomplete follow-ups

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of patients complaining of lacrimation, with subsequent detection and extraction of a dacryolit.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 1994-01; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
The percentage of individual types of amino-acids in the dacryolits | 18 months
  The obtained dacryolist were assessed physically and chemically. The authors will assess the obtained material for the presence of common amino acids.

SECONDARY OUTCOMES:
The percentage individual elements in the dacryolits | 18 months
  The obtained biological material will be assessed as regards to its elemental composition.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Kominek, doc,MD,PhD,MBA, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iliadelis ED, Karabatakis VE, Sofoniou MK. Dacryoliths in a series of dacryocystorhinostomies: histologic and chemical analysis. Eur J Ophthalmol. 2006 Sep-Oct;16(5):657-62. PMID 17061214
- [Background] Iliadelis E, Karabatakis V, Sofoniou M. Dacryoliths in chronic dacryocystitis and their composition (spectrophotometric analysis). Eur J Ophthalmol. 1999 Oct-Dec;9(4):266-8. doi: 10.1177/112067219900900402. PMID 10651189
- [Background] Lew H, Lee SY, Yun YS. Measurement of pH, electrolytes and electrophoretic studies of tear proteins in tears of patients with dacryoliths: a novel concept for dacryoliths. Ophthalmologica. 2004 Mar-Apr;218(2):130-5. doi: 10.1159/000076149. PMID 15004503
- [Derived] Kominek P, Doskarova S, Svagera Z, Lach K, Cervenka S, Zelenik K, Matousek P. Lacrimal sac dacryoliths (86 samples): chemical and mineralogic analyses. Graefes Arch Clin Exp Ophthalmol. 2014 Mar;252(3):523-9. doi: 10.1007/s00417-013-2501-6. Epub 2013 Oct 30. PMID 24170283